CLINICAL TRIAL: NCT03079258
Title: Can Physical Activity During Pregnancy Improve Maternal and Offspring Vascular Health?
Brief Title: Physical Activity and Vascular Health During Pregnancy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Liverpool John Moores University (Other)
Collaborators: Liverpool Women's NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Áine Brislane, Principal Investigator Áine Brislane, Liverpool John Moores University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 17/NW/0056
Record Dates: First submitted 2017-02-28; First posted 2017-03-14 (Actual); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Pregnant; Sedentary Lifestyle
Keywords: vascular structure; vascular function; cerebrovascular reactivity; physical activity; sedentary behaviour; offspring health; maternal health
MeSH Terms: conditions — Sedentary Behavior; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: This study comprises of two groups; an exercise and a control group.
Who Masked: Outcomes Assessor
Masking Description: Collected data at each time point will be blinded to the outcome assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): Participants randomized to the exercise intervention group will be required to complete a 24-wk partially supervised exercise programme consisting of 3-4 sessions per week of 15 minutes progressing to 30 minutes over time.
  Interventions: Other: Exercise
- Control (No Intervention): Those randomized to the control group will continue with their standard care.

INTERVENTIONS:
Other: Exercise — Previously inactive pregnant women will be asked to complete 3-4 sessions of aerobic exercise each week for 24 weeks of 15-30 minutes in duration.
  Arms: Exercise

SUMMARY:
The aim of this study is to determine the effect of aerobic exercise on maternal and offspring vascular health.

DETAILED DESCRIPTION:
The study will comprise of a randomised pilot trial to assess the effect of a moderate intensity exercise intervention on maternal and offspring vascular health. Participants will be recruited in the first trimester (T1, 10-12 weeks' gestation), and will be randomized to either a 24-week, structured and partially supervised, gym-based exercise intervention beginning in trimester 2 (T2) through to trimester 3 (T3), or a non-exercise control group who receive normal clinical care. The inclusion of this non-exercise control group is critical in allowing us to create an understanding of the adaptation of the vascular system during a normal (non-exercising) pregnancy, and also determining the physical activity and sedentary behaviour engaged in during normal healthy pregnancy. All participants will be asked to attend the laboratory at Liverpool John Moores University on 4 separate occasions synchronised with the end point of each trimester and then within four weeks of delivery. Maternal vascular health, physical activity, sedentary behaviour and fitness will be assessed during each time point throughout pregnancy while the fourth visit will comprise of an offspring vascular assessment. The investigators will also gain information on delivery outcomes including pre-term delivery, complications during labour, induction of labour, caesarean sections and post-partum haemorrhage via medical notes at the Liverpool Women's NHS Foundation Trust.

ELIGIBILITY:
Inclusion Criteria:

* Healthy pregnant female
* No history of cardiovascular disease, gestational diabetes or pre-eclampsia
* Single gestation
* Not on medication affecting cardiovascular health
* A non-smoker for at least 6 months
* Participating in structured exercise <twice/week
* BMI <30kg/m^2 -

Exclusion Criteria:

* Royal College of Obstetricians and Gynaecologists (RCOG) contraindications for pregnancy
* Pregnant by in-vitro fertilisation (IVF)exercise
* BMI >30kg/m^2
* >45 years old
* Structured exercise >twice/week
* Multiple gestation
* Disability preventing ambulation
* Currently smoking or smoking within past 6 months prior to pregnancy
* Non-English speaking women

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Due to the topic of this study, this study targets female gender.
Enrollment: 20 (Estimated)
Dates: Start 2017-04-23 (Actual); Primary Completion 2019-05-30 (Estimated); Study Completion 2019-08-03 (Estimated)

PRIMARY OUTCOMES:
Change in Vascular Function | Change from baseline at week 24 and 36 of pregnancy
  Vascular function will be measured via endothelial-dependent flow-mediated dilation (FMD) of the brachial and femoral arteries and reported as percentage change.

SECONDARY OUTCOMES:
Change in Sedentary behaviour | Change from baseline at week 24 and 36 of pregnancy
  Sedentary behaviour will be measured using an inclinometer at the end of each trimester for a period of 7 days in line with the accelerometer monitoring and will be reported in minutes.
Change in Physical activity | Change from baseline at week 24 and 36 of pregnancy
  Physical activity will be monitored for a period of 7 days using accelerometry at the end of each trimester.
Incidence of Pregnancy specific outcomes | Following delivery and within 4 weeks
  Following delivery the investigator will obtain information regarding pregnancy specific outcomes including pre-term birth, delivery complications, induction of labour, caesarean section and post-partum haemorrhage via medical notes at the collaborating hospital.

OTHER OUTCOMES:
Offspring Vascular Structure | Assessed within 4 weeks of delivery
  Offspring vascular structure will be assessed at the abdominal aorta site using ultrasound imaging. Wall thickness will be measured at three different angles of an optimised ultrasound image. The image will be adjusted so that artery wall thickness can be clearly seen and a 30 second recording taken at three different angles. The average of the three angles will be calculated for each artery. Results will be reported as change in millimetres at each time point for each artery assessed.
Change in Cerebrovascular Function | Change from baseline at week 24 and 36 of pregnancy
  Change in cerebrovascular function will be assessed using transcranial Doppler ultrasound to measure brain blood flow velocity.
Change in Vascular Structure | Change from baseline at week 24 and 36 of pregnancy
  Vascular structure will be measured at carotid, femoral and brachial arteries using ultrasound imaging to clearly visualise the artery. The image will be adjusted so that artery wall thickness can be clearly seen and a 30 second recording taken at three different angles. The average of the three angles will be calculated for each artery. Results will be reported as change in millimetres at each time point for each artery assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Hopkins, PhD, Study Director — Dr.
Locations (1):
- Research Institute for Sport and Exercise Sciences (RISES), Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brislane A, Jones H, Holder SM, Low DA, Hopkins ND. The Effect of Exercise During Pregnancy on Maternal and Offspring Vascular Outcomes: a Pilot Study. Reprod Sci. 2021 Feb;28(2):510-523. doi: 10.1007/s43032-020-00302-7. Epub 2020 Nov 30. PMID 33258064